CLINICAL TRIAL: NCT04388280
Title: Functional and Anatomic Imaging Versus No Testing in Asymptomatic High-risk Diabetic Patients
Brief Title: Imaging vs. no Testing in Asymptomatic High-risk Diabetic Patients
Acronym: FIND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Branko Beleslin, Clinical research, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 485/20
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Asymptomatic; High Risk; Diabetes
Keywords: Imaging; MACE; High risk; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Echocardiography; Global Longitudinal Strain; Computed Tomography Angiography

STUDY DESIGN:
Intervention Model Description: multi-center prospective, randomized, open label, parallel group comparison of 2 diagnostic strategies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imaging (Other): Echocardiography combined with coronary flow reserve (CFR) and strain imaging, or computed tomography (CT) angiography with direct visualization of coronary arteries.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: CT angiography
- Observation (No Intervention): No imaging for the estimation of coronary artery disease

INTERVENTIONS:
Diagnostic Test: Echocardiography — Functional assessment of coronary artery disease
  Other Names: Coronary flow reserve (CFR); Wall motion abnormalities (WMA); Strain
  Arms: Imaging
Diagnostic Test: CT angiography — Anatomical assessment of coronary artery disease
  Arms: Imaging

SUMMARY:
The aim of our study was to evaluate 1- and 3-year outcome of alternative imaging strategies in asymptomatic high-risk diabetic patients: functional stress echocardiography combined with coronary flow reserve (CFR) and strain imaging, or computed tomography (CT) angiography with direct visualization of coronary arteries, and no testing at all.

DETAILED DESCRIPTION:
A meta-analysis of >100 prospective studies, showed that diabetes mellitus (DM) in general carries a two-fold excess risk of vascular outcomes (coronary artery disease, ischemic stroke, and vascular deaths), independent of other risk factors (1). Although type 2 diabetes mellitus (DM) is far more common than type 1 DM, these results confirm adverse prognosis in both populations, which is particularly severe in the young in general and young onset female individuals with type 1 DM, emphasizing the need for intensive risk-factor management in these groups.

According to new 2019 European Society of Cardiology (ESC) / European Association for the study of diabetes (EASD) guidelines for diabetes, pre-diabetes and cardiovascular diseases (2) individuals with DM and cardiovascular diseases (CVD), or DM with target organ damage, such as proteinuria or renal failure (estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2), are at very high risk (10-year risk of CVD death >10%). Patients with DM with three or more major risk factors, or with a DM duration of >20 years, are also at very high risk. Type 1 DM at the age of 40 years with early onset (i.e. 1-10 years of age) and particularly female are associated with very high CV risk (2). Most others with DM are high risk, 10 year risk of cardiovascular diseases death (CVD) 5-10%, with the exception of young patients (aged <35 years) with type 1 DM of short duration (<10 years), and patients with type 2 DM aged <50 years with a DM duration of <10 years and without major risk factors, who are at moderate risk.

Screening for asymptomatic CAD in patients with DM remains controversial. According to current guidelines only resting ECG is recommended in patients with suspected CVD, whereas computed tomography (CT) angiography or functional imaging (radionuclide myocardial perfusion imaging, magnetic resonance imaging, or physical or pharmacological stress echocardiography) may be considered (class IIb) in asymptomatic patients with DM for screening of coronary artery disease (CAD) (2). With CT, non-invasive estimation of the atherosclerotic burden (based on the coronary artery calcium score) and identification of atherosclerotic plaques causing significant coronary stenosis (CT angiography) can be performed. Patients with DM have a higher prevalence of coronary artery calcification compared with age- and sex-matched subjects without DM (3). While a coronary artery calcium (CAC) score of 0 is associated with favorable prognosis in asymptomatic subjects with DM, each increment in CAC score (from 1 - 99 to 100 - 399 and ≥400) is associated with a 25 - 33% higher relative risk of mortality (3). Importantly, CAC is not always associated with ischemia. Therefore, coronary artery calcium score may be considered as risk modifier in CV assessment in asymptomatic patients with moderate risk (2).

Stress testing with myocardial perfusion imaging or stress echocardiography allows the detection of myocardial ischemia, particularly silent form which is more prevalent in patients with DM as demonstrated by observational studies (22%) (4-6). Randomized trials evaluating the impact of routine screening for CAD in asymptomatic DM and no history of CAD have shown no differences in cardiac death and unstable angina at follow-up in those who underwent stress testing, or CT angiography (4,6,7). A meta-analysis of five randomized studies with 3299 asymptomatic subjects with DM showed that non-invasive imaging for CAD did not significantly reduce event rates of non-fatal myocardial infarction (MI) (relative risk 0.65; P=0.062) and hospitalization for heart failure (HF) (relative risk 0.61;P=0.1) (8).Observed low event rates in these studies and the disparities in patient population and the management of screening results (different imaging techniques, invasive coronary angiography and revascularization were not performed systematically) may explain the lack of benefit of the screening strategy. Accordingly, routine screening of CAD in asymptomatic DM is not recommended (2, 8) However, stress testing or CT angiography may be indicated in very high-risk asymptomatic individuals (with peripheral arterial disease (PAD), a high CAC score, proteinuria, or renal failure) (9).

The addition of circulating biomarkers for CV risk assessment has limited clinical value (10). In patients with DM without known CVD, measurement of C-reactive protein or fibrinogen (inflammatory markers) provides minor incremental value to current risk assessment. The addition of hs troponin (Tn) T to conventional risk factors has not shown incremental discriminative power in this group (11). In individuals with type 1 DM, elevated high sensitive troponin T (hsTnT) was an independent predictor of renal decline and CV events (12). The prognostic value of N-terminal pro-B-type natriuretic peptide (NT-pro BNP) in an unselected cohort of people with DM (including known CVD) showed that patients with low levels of NT-pro BNP (<125 pg/mL) have an excellent short-term prognosis (13).

With emerging role of CT angiography in diagnosis of CAD according to the last 2019 ESC guidelines on Chronic coronary syndrome (14), as well as advanced functional imaging techniques, there is an obvious gap in evidence on prognostic value of both functional and angiographic advanced imaging techniques in patients with diabetes, particularly high risk subgroup.

The investigators hypothesized that a strategy using either functional evaluation with advanced stress echocardiography using wall motion abnormalities, coronary flow reserve and strain, or CT angiography visualization will lead to better outcome than no testing at all in asymptomatic high risk diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic patients (>30 years) with duration of diabetes ≥10 years without target organ damage plus any other additional risk factor including age, hypertension, dyslipidemia, smoking, and obesity.

Exclusion Criteria:

* Patient categorized as very high or moderate risk for CV diseases
* Any symptoms suggestive of angina or heart failure
* Patients with baseline ECG or echo abnormalities
* Patients with known CV disease, or previous myocardial revascularization
* Patients with target organ damage defined as proteinuria, renal impairment defined as eGFR <30 mL/min/1.73 m2, left ventricular hypertrophy, or retinopathy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 1 to 3 years
  Number of participants with all-cause mortality, non-fatal MI and unstable angina

SECONDARY OUTCOMES:
Individual MACE | 1 to 3 years
  Number of participants with all-cause mortality, cardiovascular mortality, non-fatal MI, revascularization (PCI or CABG), acute coronary syndrome, appearance and/or hospitalization for angina, and stroke
Testing-driven invasive angiography and revascularization | 1 to 3 years
  Number of participants undergoing invasive coronary angiography (ICA) and revascularization and rate of MACE due to invasive angiogaphy and revascularization
Prognostic role of iFR/FFR imaging in patients referred to angiography | 1 to 3 years
  Number of participants with MACE and rate of MACE in patients undergoing instantaneous wave-free ratio (iFR) and fractional flow reserve in (FFR)
Safety and outcome of revascularization in testing arms | 1 to 3 years
  Number of participants with MACE and rate of MACE due to revascularization
The role of biomarkers in high risk DM patients on their outcome (MACE) | 1 to 3 years
  Value of C-reactive protein (CRP), NT-pro BNP, and hsTnT in all participants
The impact of antidiabetic therapy and sugar control in high risk DM patients on their outcome | 1 to 3 years
  Number of participants with MACE and rate of MACE in high risk DM participants regarding antidiabetic therapy
Differences in the outcome between functional and angiographic imaging in imaging arm | 1 to 3 years
  Number of participants with MACE and rate of MACE regarding the initial imaging modality

CONTACTS AND LOCATIONS:
Overall Officials: Branko Beleslin, MD, PhD, Principal Investigator — Clinical Centre of Serbia; Nebojsa Lalic, MD, PhD, Principal Investigator — Clinical Centre of Serbia; Milos Zarkovic, MD, PhD, Principal Investigator — Clinical Centre of Serbia
Locations (1):
- Clinical Centre of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Result] Cosentino F, Grant PJ, Aboyans V, Bailey CJ, Ceriello A, Delgado V, Federici M, Filippatos G, Grobbee DE, Hansen TB, Huikuri HV, Johansson I, Juni P, Lettino M, Marx N, Mellbin LG, Ostgren CJ, Rocca B, Roffi M, Sattar N, Seferovic PM, Sousa-Uva M, Valensi P, Wheeler DC; ESC Scientific Document Group. 2019 ESC Guidelines on diabetes, pre-diabetes, and cardiovascular diseases developed in collaboration with the EASD. Eur Heart J. 2020 Jan 7;41(2):255-323. doi: 10.1093/eurheartj/ehz486. No abstract available. PMID 31497854
- [Result] Valenti V, Hartaigh BO, Cho I, Schulman-Marcus J, Gransar H, Heo R, Truong QA, Shaw LJ, Knapper J, Kelkar AA, Sciarretta S, Chang HJ, Callister TQ, Min JK. Absence of Coronary Artery Calcium Identifies Asymptomatic Diabetic Individuals at Low Near-Term But Not Long-Term Risk of Mortality: A 15-Year Follow-Up Study of 9715 Patients. Circ Cardiovasc Imaging. 2016 Feb;9(2):e003528. doi: 10.1161/CIRCIMAGING.115.003528. PMID 26848062
- [Result] Wackers FJ, Young LH, Inzucchi SE, Chyun DA, Davey JA, Barrett EJ, Taillefer R, Wittlin SD, Heller GV, Filipchuk N, Engel S, Ratner RE, Iskandrian AE; Detection of Ischemia in Asymptomatic Diabetics Investigators. Detection of silent myocardial ischemia in asymptomatic diabetic subjects: the DIAD study. Diabetes Care. 2004 Aug;27(8):1954-61. doi: 10.2337/diacare.27.8.1954. PMID 15277423
- [Result] Zellweger MJ, Maraun M, Osterhues HH, Keller U, Muller-Brand J, Jeger R, Pfister O, Burkard T, Eckstein F, von Felten S, Osswald S, Pfisterer M. Progression to overt or silent CAD in asymptomatic patients with diabetes mellitus at high coronary risk: main findings of the prospective multicenter BARDOT trial with a pilot randomized treatment substudy. JACC Cardiovasc Imaging. 2014 Oct;7(10):1001-10. doi: 10.1016/j.jcmg.2014.07.010. Epub 2014 Sep 17. PMID 25240454
- [Result] Lievre MM, Moulin P, Thivolet C, Rodier M, Rigalleau V, Penfornis A, Pradignac A, Ovize M; DYNAMIT investigators. Detection of silent myocardial ischemia in asymptomatic patients with diabetes: results of a randomized trial and meta-analysis assessing the effectiveness of systematic screening. Trials. 2011 Jan 26;12:23. doi: 10.1186/1745-6215-12-23. PMID 21269454
- [Result] Young LH, Wackers FJ, Chyun DA, Davey JA, Barrett EJ, Taillefer R, Heller GV, Iskandrian AE, Wittlin SD, Filipchuk N, Ratner RE, Inzucchi SE; DIAD Investigators. Cardiac outcomes after screening for asymptomatic coronary artery disease in patients with type 2 diabetes: the DIAD study: a randomized controlled trial. JAMA. 2009 Apr 15;301(15):1547-55. doi: 10.1001/jama.2009.476. PMID 19366774
- [Result] Clerc OF, Fuchs TA, Stehli J, Benz DC, Grani C, Messerli M, Giannopoulos AA, Buechel RR, Luscher TF, Pazhenkottil AP, Kaufmann PA, Gaemperli O. Non-invasive screening for coronary artery disease in asymptomatic diabetic patients: a systematic review and meta-analysis of randomised controlled trials. Eur Heart J Cardiovasc Imaging. 2018 Aug 1;19(8):838-846. doi: 10.1093/ehjci/jey014. PMID 29452348
- [Result] Authors/Task Force Members; Ryden L, Grant PJ, Anker SD, Berne C, Cosentino F, Danchin N, Deaton C, Escaned J, Hammes HP, Huikuri H, Marre M, Marx N, Mellbin L, Ostergren J, Patrono C, Seferovic P, Uva MS, Taskinen MR, Tendera M, Tuomilehto J, Valensi P, Zamorano JL; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; De Backer G, Sirnes PA, Ezquerra EA, Avogaro A, Badimon L, Baranova E, Baumgartner H, Betteridge J, Ceriello A, Fagard R, Funck-Brentano C, Gulba DC, Hasdai D, Hoes AW, Kjekshus JK, Knuuti J, Kolh P, Lev E, Mueller C, Neyses L, Nilsson PM, Perk J, Ponikowski P, Reiner Z, Sattar N, Schachinger V, Scheen A, Schirmer H, Stromberg A, Sudzhaeva S, Tamargo JL, Viigimaa M, Vlachopoulos C, Xuereb RG. ESC Guidelines on diabetes, pre-diabetes, and cardiovascular diseases developed in collaboration with the EASD: the Task Force on diabetes, pre-diabetes, and cardiovascular diseases of the European Society of Cardiology (ESC) and developed in collaboration with the European Association for the Study of Diabetes (EASD). Eur Heart J. 2013 Oct;34(39):3035-87. doi: 10.1093/eurheartj/eht108. Epub 2013 Aug 30. No abstract available. PMID 23996285
- [Result] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Result] Price AH, Weir CJ, Welsh P, McLachlan S, Strachan MWJ, Sattar N, Price JF. Comparison of non-traditional biomarkers, and combinations of biomarkers, for vascular risk prediction in people with type 2 diabetes: The Edinburgh Type 2 Diabetes Study. Atherosclerosis. 2017 Sep;264:67-73. doi: 10.1016/j.atherosclerosis.2017.07.009. Epub 2017 Jul 12. PMID 28777936
- [Result] Galsgaard J, Persson F, Hansen TW, Jorsal A, Tarnow L, Parving HH, Rossing P. Plasma high-sensitivity troponin T predicts end-stage renal disease and cardiovascular and all-cause mortality in patients with type 1 diabetes and diabetic nephropathy. Kidney Int. 2017 Nov;92(5):1242-1248. doi: 10.1016/j.kint.2017.04.018. Epub 2017 Jul 14. PMID 28712855
- [Result] Huelsmann M, Neuhold S, Strunk G, Moertl D, Berger R, Prager R, Abrahamian H, Riedl M, Pacher R, Luger A, Clodi M. NT-proBNP has a high negative predictive value to rule-out short-term cardiovascular events in patients with diabetes mellitus. Eur Heart J. 2008 Sep;29(18):2259-64. doi: 10.1093/eurheartj/ehn334. Epub 2008 Jul 23. PMID 18650200
- [Result] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- See also: Chow S, Shao J, Wand H. Sample size calculations in clinical research. 2nd edition. 2008. — https://www.mobt3ath.com/uplode/book/book-43792.pdf